CLINICAL TRIAL: NCT06457152
Title: Multi-Center Project: BETTER CARE - HF (Building Electronic Tools To Enhance and Reinforce CArdiovascular REcommendations - Heart Failure)
Brief Title: Multi-Center Project: Building Electronic Tools To Enhance and Reinforce CArdiovascular REcommendations - Heart Failure
Acronym: BETTER CARE-HF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Massachusetts General Hospital (Other); University of Pennsylvania (Other); OhioHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-00179
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants who are randomized to receive the intervention (i.e., displaying the automated EHR-embedded alert).
  Interventions: Other: EHR-Emedded Alert
- Standard of Care (No Intervention): Participants who are randomized to the control group (i.e., not displaying the automated EHR-embedded alert).

INTERVENTIONS:
Other: EHR-Emedded Alert — For patients randomized to the intervention group, an automated, EHR-embedded alert will be visible in the patient's chart that promotes appropriate medical therapy for patients with HFrEF.
  Arms: Intervention

SUMMARY:
This study will test an automated, electronic health record (EHR-)embedded alert to improve prescribing of guideline-directed medical therapy for patients with heart failure and reduced ejection fraction (HFrEF). The investigators have previously tested and implemented this alert at NYU Langone Health (NYULH), and will now test and implement this alert across three other health systems.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an encounter visit at participating cardiology practice during the study period
* Patient with EF of less than or equal to 40% on most recent echocardiogram at the time of visit
* Patient ages 18-90

Exclusion Criteria:

* Pregnancy
* Ventricular assist device
* Hospice
* Cardiac amyloid
* Medication-specific exclusion for MRA: most recent systolic blood pressure less than 105 mm Hg, most recent potassium < 5.1, any potassium > 5.5, most recent glomerular filtration rate < 30 (using MDRD equation), or a documented MRA allergy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2025-12-04 (Actual); Study Completion 2026-03-29 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with a Prescription for Mineralocorticoid Antagonists (MRA) | Up to Day 30
  Measured at the prescription encounter level using patient EHR data.

SECONDARY OUTCOMES:
Number of Patients with a Prescription for Beta-Blocker (BB) | Up to Day 30
  Measured at the prescription encounter level using patient EHR data.
Number of Patients with a Prescription for ACE-I/ARB/ARNI | Up to Month 36
  Prescription for angiotensin converting enzyme-inhibitors/angiotensin receptor blockers/angiotensin receptor neprilysin inhibitors (ACE-I/ARB/ARNI) measured at the prescription encounter level using patient EHR data.
Number of Patients with a Prescription for Sodium-Glucose Cotransporter-2 Inhibitor (SGLT2i) | Up to Month 36
  Measured at the prescription encounter level using patient EHR data.
Number of Patients with Hyperkalemia | Up to Month 36
  Measured using patient EHR data.
Number of Patients who are Hospitalized | Up to Month 36
  Measured using patient EHR data.
Number of Patients who are Hospitalized for Heart Failure (HF) | Up to Month 36
  Measured using patient EHR data.

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Mukhopadhyay, Principal Investigator — NYU Langone Health
Locations (4):
- United States (4):
  - University of Massachusetts, Boston, Massachusetts
  - NYU Langone Health, New York, New York
  - OhioHealth, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: amrita.mukhopadhyay@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to amrita.mukhopadhyay@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.